CLINICAL TRIAL: NCT06192706
Title: Clinical Investigation for the Foldax Tria Aortic Heart Valve India
Brief Title: Clinical Investigation for the Foldax Tria Aortic Heart Valve- India
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foldax, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Foldax CP-003
Record Dates: First submitted 2023-12-07; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency; Aortic Valve Calcification; Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Aortic Valve, Calcification of; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tria Aortic Valve (Experimental): Patients receiving the Foldax Aortic Valve
  Interventions: Device: Foldax Tria Aortic Valve

INTERVENTIONS:
Device: Foldax Tria Aortic Valve — Aortic Valve Replacement

SUMMARY:
The purpose of this study is to conduct a clinical investigation of the Foldax Tria Aortic Valve to collect evidence on the device's safety and performance.

DETAILED DESCRIPTION:
The Foldax Tria Aortic Heart Valve is indicated as a replacement for diseased, damaged, or malfunctioning native aortic heart valve via open heart surgery. The study is a single open are label non-randomized multi- center clinical trial. Up to 10 sites in the country of India will enroll up to 50 patients. These patients will follow the study schedule for 1 year after implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Is 45 years or older
2. Provide written informed consent prior to trial procedures after standard of care studies and tests indicate that the patient needs aortic valve replacement
3. Agrees to attend all follow-up assessments for up to 1 year and is willing to comply with specified follow-up evaluations for the FOLDAX Clinical trial
4. Diagnosed with symptomatic aortic valve disease (stenosis and/or regurgitation) where aortic valve replacement is recommended based on pre-operative evaluations

Exclusion Criteria:

1. Requires multiple valve replacement / repair
2. Requires emergency surgery
3. Has had prior valve surgery
4. Requires a surgical procedure outside of the cardiac area
5. Requires a cardiac procedure other than a CABG or root enlargement
6. Requires or are planning another unrelated surgery within 12 months of undergoing implantation of the study device
7. Has active endocarditis/myocarditis or within 3 months to the scheduled surgery
8. Has renal insufficiency as determined by creatinine (S-Cr) level as ≥ 1.5 mg/dl or endstage renal disease requiring chronic dialysis at screening visit
9. Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months (90 days) prior to planned valve surgery
10. Has acute myocardial infarction (Ml) within 30 days prior to planned valve surgery
11. Has life expectancy to less than 12 months
12. Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM), except patients who have isolated subaortic muscular hypertrophy diagnosed at the time of surgery
13. Diagnosed with abnormal calcium metabolism and/or hyperparathyroidism
14. Echocardiographic left ventricular ejection fraction <25%
15. Echocardiographic evidence of an intra-cardiac thrombus or vegetation
16. Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery
17. Documented leukopenia (WBC < 4.0 x 103/µL), acute anemia (Hgb < 10.0 gm/dl or 6 mmol/L), thrombocytopenia (platelet count < 100 x103/µL) or history of bleeding diathesis or coagulopathy
18. Has prior organ transplant or is currently an organ transplant candidate
19. Current or recent participation (within 6 weeks prior to surgery) in another drug or device trial
20. Pregnant, lactating or planning to become pregnant during the duration of participation in trial
21. Currently incarcerated or unable to give voluntary informed consent
22. Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant
23. Requires concomitant left ventricular assist device (LVAD) placement, Impella placement, and/or intra-aortic balloon pump
24. Tests positive for an active infection with SARS-CoV-2 (COVID-19)
25. Currently diagnosed as uncontrolled diabetes mellitus (Random BLS > 300 mg/dl)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints: Clinical Outcomes Event Assessment | 12 months following patient enrollment completion
  The rate of adverse events will be compared to clinical outcomes for surgically implanted heart valves reported in the literature: a) thromboembolism, b) valve thrombosis, c) major paravalvular leak, d) major hemorrhage, e) endocarditis, f) all-caused death, g) valve related death, h) valve related reoperation, i) valve explant, j) hemorrhage, k) all-cause reoperation
Primary Effectiveness Endpoint: Hemodynamic Performance Assessment | 12 months following patient enrollment completion
  Hemodynamic performance parameters are mmHG mean gradient and derived Effective Orifice Area (EOA). Success is defined as clinically significant improvement in hemodynamic performance (Effective Orifice Area (EOA)) at one year based on literature reports for surgical aortic valve replacement.
Primary Effectiveness Endpoint: New York Heart Association Improvement Assessment | 12 months following patient enrollment completion
  Clinically significant improvement (one grade) in the New York Heart Association (NYHA) functional classification status at 365 days compared to baseline. a. Class I - No symptoms and no limitations in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. b. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. c. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100m). Comfortable only at rest. d. Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

SECONDARY OUTCOMES:
Stroke | 12 months following patient enrollment
  Assessment of patient experiencing a stroke verified by imaging and or physical exam
Transient Ischemic Attack | 12 months following patient enrollment
  Assessment of patient having a TIA verified by imaging and or physical exam
ICU Duration of Stay | 30 days post procedure
  Length of stay in the ICU post valve implantation defined as arrival time/date in hours and minutes to transfer to floor time/date in hours and minutes.
Ventilation Time | 30 Days post procedure
  Ventilation time in hours defined as arrival time/date in recovery in hours and minutes to date and time extubated in hours and minutes
New Onset Atrial Fibrillation | 12 Months post procedure
  New/post-operative atrial fibrillation - confirmed on ECG after closure during initial or subsequent admission or at one-year review
Length of Stay in Hospital | 30 Days post procedure
  Post procedure length of stay defined as the date and time in hours and minutes documented for arrival in the recovery unit to date and time in hours and minutes of discharge in hours and minutes.
Readmission | 30 Days post procedure
  Patient readmission to the hospital post discharge measured by date/time
Hemolysis screen | 12 Months post procedure
  Hemolysis screen is measured by blood tests including hemoglobin and liver enzyme assessments
Change in Quality of Life (QOL) | 12 Months post procedure
  Change in QOL as measured by the Kansas City Cardiomyopathy Questionnaire
Six Minute Walk Test (6MWT) | 12 months post procedure
  Change in distance walked during a 6MWT

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal Pandey, MBBS, MS, Principal Investigator — Hinduja Hospital
Locations (10):
- India (10):
  - GCS Medical College, Ahmedabad, Gujarat
  - Epic Hospital, Ahmedabad, Gujarat
  - KEM Hospital, Mumbai, Maharashtra
  - Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Six Sigma, Nashik, Maharashtra
  - B.J. Medical College, Pune, Maharashtra
  - SMS Hospital, Jaipur, Rajasthan
  - Indo-US Hospital, Hyderabad, Telangana
  - NRS Medical College and Hospital, Kolkata, West Bengal
  - Fortis Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No